CLINICAL TRIAL: NCT04499651
Title: Adaptation and Testing of a Navigation Intervention for Hepatitis C and HIV Co-infected Persons Leaving LA County Jail
Brief Title: Testing of a Navigation Intervention for Hepatitis C and HIV
Acronym: LINKHCV
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient enrollment numbers due to Covid-19 pandemic
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, David Goodman-Meza, MD, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: ISR-US-18-10586
Record Dates: First submitted 2020-07-28; First posted 2020-08-05 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: HIV (Human Immunodeficiency Virus); Hepatitis C
Keywords: HIV; Hepatitis C; Corrections; Engagement-in-care; Navigation; Criminal justice system
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Hepatitis C

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): All people who are living with HIV who are currently in custody in the Los Angeles County Jail are provided with Transitional Case Management and may also receive Whole Person Care related services regardless of participation in this study. Participants recruited from clinics who do not enroll in the study will be offered HIV/HCV care that follows the national HIV/HCV care guidelines, as provided by participating study clinics. Participants recruited from non-medical community agencies who do not enroll in the study and do not have a regular provider will receive a referral list of HIV/HCV care facilities that follow the national HIV/HCV care guidelines.
- Navigation (Active Comparator): Participants will be paired with a navigator and will complete the following didactic sessions in one-on-one format:
  1. Session 1: Intervention Overview and Basic HIV/HCV Knowledge and Skills Builder
  2. Session 2: Rapport Building
  3. Session 3: Society and Self and the Role of Disclosure
  4. Session 4: Accompaniment 1
  5. Session 5: Goal-Setting, Problem-Solving and a Disclosure Toolkit
  6. Session 6: Accompaniment 2
  7. Session 7: Accompaniment 3 (ONLY if needed)
  8. Weekly check-in calls following Session 2 for six months
  Interventions: Behavioral: Navigation

INTERVENTIONS:
Behavioral: Navigation — Trained study navigators will provide one-on-one learning sessions and accompaniments to criminal-justice involved people to help link them to HIV/Hepatitis C care
  Arms: Navigation

SUMMARY:
This study will evaluate the efficacy of navigation for hepatitis C treatment in people living with both HIV and HCV with criminal justice involvement.

DETAILED DESCRIPTION:
Hepatitis C (HCV) is the most common chronic, blood-borne infection in the U.S. and, untreated, can result in liver failure and liver cancer. Despite advances in treatment and remarkable improvements in cure rates, very few persons with chronic HCV infection are receiving this treatment, especially among people who use drugs, who are also disproportionately HIV-infected and incarcerated. Existing efforts to ensure linkage to and retention in medical care following release from incarceration among people living with both HIV and HCV are generally insufficient. Increasing treatment engagement following release from incarceration can drastically reduce HCV and HIV in the blood, which can limit transmission to sexual and injection drug use partners.

The goal of this study is to evaluate the effect of a novel navigation intervention to improve HIV/HCV treatment engagement among HIV/HCV co-infected adults with criminal justice involvement. The investigators hypothesize that the navigation intervention is more effective than the current standard-of-care approaches to link this population of adults to HIV/HCV treatment. All participants, regardless of study arm, will complete one baseline interview around the time of study enrollment. Follow-up interviews are done at 3 months and 8 months following enrollment (if enrolled in the community) or after release from jail (if enrolled in the jail).

Blood samples to analyze the HCV RNA will be collected or requested from participants' clinics both for the baseline assessment and the assessment conducted 12 weeks after completion of the HCV treatment course (if the HCV RNA result cannot be obtained at 12 weeks, it will done at the 8-month follow-up interview). HIV RNA will be collected from the clinics.

In addition to the interviews and the HCV/HIV RNA assessments, participants assigned to the intervention arm will engage in a six- or seven-session navigation intervention. Participants will be in the study for about 12 months but no more than 3 years.

ELIGIBILITY:
Inclusion Criteria (if recruited in jail)

1. Diagnosed HIV+/HCV co-infection;
2. 18 years of age or older;
3. non-cis women;
4. Fluent in speaking English;
5. Have an anticipated sentence of no more than 12 months;
6. Have detectable Hepatitis C viral load
7. Going to live in LA County, Kern County, San Diego County, Riverside County, Ventura County or San Bernardino County

If recruited outside of jail:

1. Diagnosed HIV+/HCV co-infection;
2. 18 years of age or older;
3. non-cis women;
4. Fluent in speaking English;
5. Incarceration history within the last 12 months of enrollment;
6. Have detectable Hepatitis C viral load
7. Going to live in LA County, Kern County, San Diego County, Riverside County, Ventura County or San Bernardino County

Exclusion Criteria:

1. Inability to give informed consent
2. CD4 count<200

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — All cis-men (assigned "male" at birth) are eligible for the study regardless of current gender identification.
Enrollment: 1 (Actual)
Dates: Start 2020-07-31 (Actual); Primary Completion 2021-02-22 (Actual); Study Completion 2021-02-22 (Actual)

PRIMARY OUTCOMES:
Undetectable Hepatitis C RNA | 8 months
  Undetectable Hepatitis C RNA
Undetectable HIV RNA | 8 months
  HIV RNA <40 copies/ml

CONTACTS AND LOCATIONS:
Overall Officials: David Goodman-Meza, MD, MAS, Principal Investigator — University of California, Los Angeles; Debika Bhattacharya, MD, MSc, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA, Los Angeles, California, United States